CLINICAL TRIAL: NCT00979212
Title: Randomized Phase II Study of Pre-operative Chemoradiotherapy +/- Panitumumab (IND #110152) Followed by Consolidation Chemotherapy in Potentially Operable Locally Advanced (Stage IIIA, N2+) Non-Small Cell Lung Cancer
Brief Title: Chemotherapy and Radiation Therapy With or Without Panitumumab in Treating Patients With Stage IIIA Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RTOG-0839; CDR0000654690; NCT00979212 (Registry Identifier: Clinical Trials.gov ID); NCI-2011-01970 (Registry Identifier: Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2009-09-16; First posted 2009-09-17 (Estimated); Results first posted 2016-08-16 (Estimated); Last update posted 2022-06-15 (Actual); Status verified 2022-05

CONDITIONS: Lung Cancer
Keywords: stage IIIA non-small cell lung cancer; adenocarcinoma of the lung; adenosquamous cell lung cancer; bronchoalveolar cell lung cancer; large cell lung cancer; squamous cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung; Adenocarcinoma, Bronchiolo-Alveolar | interventions — Panitumumab; Carboplatin; Paclitaxel; Albumin-Bound Paclitaxel; Surgical Procedures, Operative; Anterior Temporal Lobectomy; Pneumonectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Induction CT+RT (Active Comparator): Chemotherapy (paclitaxel and carboplatin) plus radiation therapy followed by surgery (if operable) followed by consolidation chemotherapy (paclitaxel and carboplatin)
  Interventions: Drug: carboplatin; Drug: paclitaxel; Procedure: surgery
- Induction CT+RT+Panitumumab (Experimental): Panitumumab plus chemotherapy (paclitaxel and carboplatin) plus radiation therapy followed by surgery (if operable) followed by consolidation chemotherapy (paclitaxel and carboplatin)
  Interventions: Drug: panitumumab; Drug: carboplatin; Drug: paclitaxel; Procedure: surgery

INTERVENTIONS:
Drug: panitumumab — Induction: 2.5 mg/kg, IV, days 1, 8, 15, 22, 29, 36 of radiation therapy before administration of chemotherapy and radiation therapy.
  Other Names: Vectibix
  Arms: Induction CT+RT+Panitumumab
Drug: carboplatin — Induction: AUC=2, IV, days 1, 8, 14, 22, 29, and 36 of radiation therapy. Consolidation, 6-12 weeks following surgery, AUC=6, IV, days 1 and 22.
  Other Names: Paraplatin
Drug: paclitaxel — Induction: 50 mg/m2, IV, days 1, 8, 14, 22, 29, and 36 of radiation therapy. Consolidation, 6-12 weeks following surgery, 200 mg/m2, IV, days 1 and 22.
  Other Names: Taxol; Abraxane
Procedure: surgery — A lobectomy or pneumonectomy performed 4-6 weeks after completion of induction chemoradiation
  Other Names: lobectomy; pneumonectomy

SUMMARY:
RATIONALE: Drugs used in chemotherapy (CT), such as paclitaxel and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy (RT) uses high-energy x-rays to kill tumor cells. Monoclonal antibodies, such as panitumumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Giving these treatments before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed. It is not yet known whether chemotherapy and radiation therapy are more effective when given with or without panitumumab in treating patients with non-small cell lung cancer.

PURPOSE: This randomized phase II trial is studying chemotherapy and radiation therapy to see how well they work when given with or without panitumumab in treating patients with stage IIIA non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the mediastinal nodal clearance after completion of induction chemoradiotherapy with or without panitumumab in patients with stage IIIA non-small cell lung cancer.

Secondary

* Assess overall survival of these patients.
* Evaluate patterns of first failure in these patients.
* Determine the acute and late adverse events associated with these regimens.
* Assess surgical morbidities in patients with resectable disease at reassessment.
* Determine the correlation between pre- and post-treatment biomarkers (including epidermal growth factor receptor (EGFR) and ras mutation status) and outcomes (mediastinal nodal clearance and overall survival).
* Evaluate the prognostic value of plasma osteopontin and microRNA for overall survival.
* Assess the ability of FDG-PET/CT scan re-staging to predict outcome.

OUTLINE: This is a multicenter study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive induction therapy comprising paclitaxel IV over 1 hour and carboplatin IV over 30 minutes on days 1, 8, 15, 22, 29, and 36. Patients also undergo intensity-modulated radiotherapy (IMRT) or 3-dimensional conformal radiotherapy (3D-CRT) once daily on days 1-5, 8-12, 15-19, 22-26, 29-33, and 36-40. Beginning approximately 6-12 weeks later, patients receive consolidation therapy comprising paclitaxel IV over 1 hour and carboplatin IV over 30 minutes on days 1 and 21.
* Arm II: Patients receive induction therapy comprising panitumumab IV over 1 hour on days 1, 8, 15, 22, 29, and 36 and paclitaxel IV over 1 hour and carboplatin IV over 30 minutes on days 8, 15, 22, 29, and 36. Patients also undergo IMRT or 3D-CRT once daily on days 8-12, 15-19, 22-26, 29-33, 36-40, and 43-47. Beginning approximately 6-12 weeks later, patients receive consolidation therapy comprising paclitaxel IV over 1 hour and carboplatin IV over 30 minutes on days 1 and 21.
* In both arms, patients with resectable disease and no disease progression may proceed to surgery (thoracotomy, lobectomy, or pneumonectomy) approximately 4-6 weeks after completion of induction therapy. After surgery, patients proceed to consolidation therapy.

After completion of study treatment, patients are followed up at 6 weeks, every 3 months for 1 year, every 6 months for 2 years, and then annually thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed* non-small cell lung cancer (NSCLC), including any of the following histologies:

  * Adenocarcinoma
  * Adenosquamous
  * Large cell carcinoma
  * Squamous cell carcinoma
  * Non-lobar and non-diffuse bronchoalveolar cell carcinoma
  * NSCLC not otherwise specified NOTE: *Documentation of NSCLC may originate from the mediastinal node biopsy or aspiration
* Stage IIIA (T1-T3) disease with a single primary lung parenchymal lesion AND positive ipsilateral mediastinal node or nodes (N2) with or without positive ipsilateral hilar nodes (N1)

  * N2 nodes must be separate from primary tumor by either CT scan or surgical exploration
  * Maximum nodal diameter of involved N2 nodes cannot exceed 3.0 cm
  * N2 status must be pathologically confirmed to be positive by one of the following methods*:

    * Mediastinoscopy
    * Mediastinotomy (Chamberlain procedure)
    * Transesophageal needle biopsy using endoscopic ultrasound (EUS-TBNA)
    * Endobronchial ultrasound biopsy using endoscopic ultrasound guidance (EBUS-TBNA)
    * Thoracotomy
    * Video-assisted thoracoscopy
    * Transbronchial needle biopsy by Wang technique (TBNA)
    * Fine-needle aspiration under CT guidance NOTE: *PET positivity in the ipsilateral mediastinal lymph nodes is not sufficient to establish N2 nodal status
  * Ipsilateral mediastinal nodes associated with right-sided tumor must be biopsied unless all of the following are true:

    * Tumor is left sided
    * Paralyzed left true vocal cord documented by bronchoscopy or indirect laryngoscopy
    * Nodes visible in the anterior/posterior (level 5) region on CT scan
    * Distinct primary tumor separate from nodes visible on CT scan
    * Histologic (biopsy) or cytologic (needle aspiration or sputum) proof of non-small cell histology from the primary tumor
  * If lymph nodes in the contralateral mediastinum and neck are visible on contrast CT scan of the chest and are > 1.0 cm in short axis or if contralateral involvement is suggested by PET scan, then the nodes must be confirmed to be negative
* Measurable disease as determined by contrast-enhanced CT scan

  * Primary lung tumor distinct from mediastinal lymph nodes
* If a pleural effusion is present, the following criteria must be met to exclude malignant involvement (incurable M1a disease):

  * When pleural fluid is visible on both the CT scan and on a chest x-ray, a pleuracentesis is required to confirm that the pleural fluid is cytologically negative.
  * Exudative pleural effusions are excluded, regardless of cytology;
  * Effusions that are minimal (i.e. not visible under ultrasound guidance) that are too small to safely tap are eligible.
* No palpable lymph nodes in the supraclavicular areas or higher in the neck, unless proven to be benign by fine-needle aspiration or biopsy
* No distant metastases

PATIENT CHARACTERISTICS:

* Zubrod performance status 0-1
* Absolute neutrophil count (ANC) ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 10.0 g/dL (transfusion allowed)
* Creatinine clearance ≥ 60 mL/min
* Total bilirubin ≤ 1.5 times upper limit of normal (ULN)
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 times ULN
* Alkaline phosphatase ≤ 2.5 times ULN
* Serum albumin > 3.0 g/dL
* Serum magnesium normal (supplementation allowed)
* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 6 months after completion of treatment
* Forced expiratory volume at one second (FEV1) ≥ 2.0 L OR predicted post-resection FEV1 ≥ 0.8 L
* Diffusion capacity ≥ 50% predicted
* No other invasive malignancy within the past 3 years, except nonmelanoma skin cancer or carcinoma in situ of the breast, oral cavity, or cervix
* No severe, active co-morbidity, including any of the following:

  * Current uncontrolled cardiac disease (e.g., uncontrolled hypertension, unstable angina, myocardial infarction within the past 6 months, uncontrolled congestive heart failure, or cardiomyopathy with decreased ejection fraction (<50%)
  * Acute bacterial or fungal infection requiring IV antibiotics
  * Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or that would preclude study therapy within the past 4 weeks
  * Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects
  * AIDS or known HIV positivity
* No unintentional weight loss ≥ 5% of body weight within the past 6 months
* No prior severe infusion reaction to a monoclonal antibody
* No pre-existing peripheral neuropathy ≥ grade 2

PRIOR CONCURRENT THERAPY:

* No prior systemic chemotherapy or biological therapy (including erlotinib hydrochloride or similar agents) for the study cancer

  * Prior chemotherapy for a different cancer allowed
* No prior radiotherapy to the region of the study cancer that would result in overlap of radiotherapy fields
* No prior therapy that specifically and directly targets the EGFR pathway

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2011-02; Primary Completion 2015-12 (Actual); Study Completion 2022-05-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin J. Edelman, MD, Principal Investigator — University of New Maryland
Locations (31):
- United States (31):
  - Mercy Cancer Center at Mercy San Juan Medical Center, Carmichael, California
  - Radiological Associates of Sacramento Medical Group, Incorporated, Sacramento, California
  - Penrose Cancer Center at Penrose Hospital, Colorado Springs, Colorado
  - Lucille P. Markey Cancer Center at University of Kentucky, Lexington, Kentucky
  - CCOP - Ochsner, New Orleans, Louisiana
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - St. Agnes Hospital Cancer Center, Baltimore, Maryland
  - Cancer Institute at St. Joseph Medical Center, Towson, Maryland
  - Boston University Cancer Research Center, Boston, Massachusetts
  - Fairview Southdale Hospital, Edina, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - Methodist Estabrook Cancer Center, Omaha, Nebraska
  - NYU Cancer Institute at New York University Medical Center, New York, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Summa Center for Cancer Care at Akron City Hospital, Akron, Ohio
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Natalie Warren Bryant Cancer Center at St. Francis Hospital, Tulsa, Oklahoma
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - Cherry Tree Cancer Center, Hanover, Pennsylvania
  - Cancer Center of Paoli Memorial Hospital, Paoli, Pennsylvania
  - Kimmel Cancer Center at Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania
  - Albert Einstein Cancer Center, Philadelphia, Pennsylvania
  - McGlinn Family Regional Cancer Center at Reading Hospital and Medical Center, Reading, Pennsylvania
  - Lankenau Cancer Center at Lankenau Hospital, Wynnewood, Pennsylvania
  - York Cancer Center at Apple Hill Medical Center, York, Pennsylvania
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin
  - Veterans Affairs Medical Center - Milwaukee, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Induction CT+RT | Induction CT+RT+Panitumumab
Started | 24 | 47
Completed | 22 (Subjects with data available for primary analysis are considered to have completed the study.) | 39 (Subjects with data available for primary analysis are considered to have completed the study.)
Not Completed | 2 | 8
Not completed — Protocol Violation | 1 | 8
Not completed — No protocol therapy received | 1 | 0

BASELINE CHARACTERISTICS:
Population: All eligible patients receiving protocol treatment
Groups:
- Total: Total of all reporting groups
Arm/Group | Induction CT+RT | Induction CT+RT+Panitumumab | Total
Number analyzed (Participants) | 22 | 39 | 61
Age, Continuous [Median (Full Range); unit: years] | 61 [51 to 77] | 61 [32 to 78] | 61 [32 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 18 | 31
  Male | 9 | 21 | 30

OUTCOME MEASURES:

1. Primary Outcome: Mediastinal Nodal Clearance After Completion of Induction Chemoradiotherapy With or Without Panitumumab.
Description: The assessment of whether mediastinal nodes which were involved at the time of study registration were clear of disease following induction chemoradiotherapy with or without panitumumab; the assessment is made at the time of surgery 4-6 weeks after chemoradiation. If surgery could not be performed, the patient was considered as not having had mediastinal nodal clearance.
Time Frame: From date of randomization to time of protocol surgery, approximately 12 weeks.
Population: All eligible patients who started study treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Induction CT+RT | Induction CT+RT+Panitumumab
Number analyzed (Participants) | 22 | 39
percentage of participants | 68.2 [45.1 to 86.1] | 48.7 [32.4 to 65.2]
Statistical Analysis 1: Comparison: Induction CT+RT vs Induction CT+RT+Panitumumab; Null hypothesis (H0) was that the experimental treatment was not effective vs the alternative hypothesis (HA) that it was. H0: OR ≤ 1 vs. HA: OR > 1, where odds ratio (OR)= [p2*(1- p1)]/ [p1*(1- p2)], p1 denotes the mediastinal clearance rate (MCR) on Induction chemoradiation; p2 denotes the MCR on Induction chemoradiation + panitumumab. Fisher's exact test was used to compare the MCRs; the 95% confidence interval was calculated using Clopper-Pearson method. 97 patients were required; Test type: Superiority or Other; p = 0.96, Fisher Exact — One-sided test at significance level of 0.05

2. Secondary Outcome: Overall Survival
Description: Survival time was calculated from the date of randomization to the date of death from any cause or the date of last follow-up. The Kaplan-Meier method was used to estimate the overall survival rates. One-year survival rates were estimated, not compared.
Time Frame: Patients are followed until death. Analysis occurs at time of primary analysis, approximately five years from start of study
Population: All eligible patients who started study treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Induction CT+RT | Induction CT+RT+Panitumumab
Number analyzed (Participants) | 22 | 39
percentage of participants | 94.4 [66.6 to 99.2] | 89.1 [73.5 to 95.8]

3. Secondary Outcome: Patterns of First Failure
Description: The first failure site will be tabulated, not compared.
Time Frame: as for outcome 2
Population: All eligible patients who started study treatment
Measure: Number; unit: participants
Arm/Group | Induction CT+RT | Induction CT+RT+Panitumumab
Number analyzed (Participants) | 22 | 39
participants
  Alive, no failure | 15 | 20
  Dead, no failure | 1 | 3
  Distant failure only | 4 | 9
  Local and distant failure | 1 | 2
  Local and regional failure | 0 | 1
  Local, regional, and distant failure | 0 | 2
  Regional failure only | 1 | 2

4. Secondary Outcome: Percentage of Patients With Grade 3 or Higher Acute and Late Adverse Events
Description: Adverse events are graded using CTCAE v3.0. Grade refers to the severity of the AE. The CTCAE v3.0 assigns Grades 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline: Grade 1 Mild AE, Grade 2 Moderate AE, Grade 3 Severe AE, Grade 4 Life-threatening or disabling AE, Grade 5 Death related to AE. Does not include surgical morbidities. An acute adverse event is defined as any grade 3 or worse toxicity occurring during protocol treatment and within 30 days from the end of protocol treatment that is possibly, probably, or definitely related to treatment. Acute adverse events are any adverse events occurring within 30 days of the end of all protocol treatment. Late adverse events are any adverse events occurring after 30 days after the end of all protocol treatment.
Time Frame: as for outcome 2
Population: All eligible patients who started study treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Induction CT+RT | Induction CT+RT+Panitumumab
Number analyzed (Participants) | 22 | 39
percentage of participants
  Acute | 81.8 [59.7 to 94.8] | 69.2 [52.4 to 83.0]
  Late | 30.3 [11.9 to 54.3] | 15.2 [5.1 to 31.9]

5. Secondary Outcome: Surgical Morbidities in Patients With Resectable Disease at Reassessment
Description: A surgical morbidity is any toxicity occurring within 30 days of protocol surgery, as evaluated using CTCAE v4.0. Rates of grade 3 and higher surgical morbidity were calculated; the rates across arms were not compared.
Time Frame: From date of surgery to 30 days following surgery.
Population: All eligible patients who started study treatment and received protocol surgery
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Induction CT+RT | Induction CT+RT+Panitumumab
Number analyzed (Participants) | 19 | 30
percentage of patients | 42.1 [20.3 to 66.5] | 20 [7.7 to 38.6]

6. Secondary Outcome: Ability of FDG-PET/CT Scan Data to Predict Outcome
Time Frame: as for outcome 2
Population: FDG-PET/CT scan data was not obtained and therefore this outcome measure cannot be reported.
Arm/Group | Induction CT+RT | Induction CT+RT+Panitumumab
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Response Rate
Description: Patients are assessed for best response to protocol treatment using the RECIST criteria. The response rate was calculated as the number of patients who have a complete response (CR) or partial response (PR) divided by the total number of analyzable patients at completion of induction chemoradiation +/- panitumumab and prior to anticipated surgery in each arm. Patients without a documented assessment are considered as not having a CR or PR. Rates are not compared across arms.
Time Frame: From date of randomization to time of protocol surgery, approximately 12 weeks.
Population: All eligible patients who started study treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Induction CT+RT | Induction CT+RT+Panitumumab
Number analyzed (Participants) | 22 | 39
percentage of participants | 77.3 [54.6 to 92.2] | 61.5 [44.6 to 76.6]

ADVERSE EVENTS:
Description: Subjects experiencing more than one of a given adverse event are counted only once for that adverse event. Note, with yearly update of adverse events, eligibility determination of one patient changed and as a result the number at risk shown for adverse events now differs from the Participant Flow table which was entered previously.
Arm/Group | Induction CT+RT | Induction CT+RT+Panitumumab
Serious Adverse Events (participants affected / at risk) | 8/22 | 20/38
Other Adverse Events (participants affected / at risk) | 22/22 | 37/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Induction CT+RT (N=22) | Induction CT+RT+Panitumumab (N=38)
Anemia (Blood and lymphatic system disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 2
Cardiac arrest (Cardiac disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 2 | 2
Dysphagia (Gastrointestinal disorders) | 0 | 1
Esophagitis (Gastrointestinal disorders) | 1 | 2
Gastritis (Gastrointestinal disorders) | 0 | 1
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 2
Rectal hemorrhage (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 2
Fatigue (General disorders) | 0 | 1
Infusion related reaction (General disorders) | 0 | 1
Anaphylaxis (Immune system disorders) | 0 | 1
Lung infection (Infections and infestations) | 2 | 5
Pleural infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 3
Skin infection (Infections and infestations) | 0 | 1
Upper respiratory infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Wound infection (Infections and infestations) | 0 | 1
Postoperative thoracic procedure complication (Injury, poisoning and procedural complications) | 0 | 1
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 | 1
Lymphocyte count decreased (Investigations) | 1 | 2
Neutrophil count decreased (Investigations) | 1 | 2
White blood cell decreased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Nervous system disorders - Other (Nervous system disorders) | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0
Recurrent laryngeal nerve palsy (Nervous system disorders) | 1 | 0
Stroke (Nervous system disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchial stricture (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchopleural fistula (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1
Thromboembolic event (Vascular disorders) | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Induction CT+RT (N=22) | Induction CT+RT+Panitumumab (N=38)
Anemia (Blood and lymphatic system disorders) | 13 | 20
Atrial fibrillation (Cardiac disorders) | 7 | 4
Atrial flutter (Cardiac disorders) | 2 | 0
Chest pain - cardiac (Cardiac disorders) | 2 | 0
Sinus tachycardia (Cardiac disorders) | 5 | 2
Ventricular arrhythmia (Cardiac disorders) | 3 | 0
Constipation (Gastrointestinal disorders) | 6 | 17
Diarrhea (Gastrointestinal disorders) | 7 | 7
Dyspepsia (Gastrointestinal disorders) | 7 | 11
Dysphagia (Gastrointestinal disorders) | 9 | 17
Esophagitis (Gastrointestinal disorders) | 8 | 15
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 | 4
Nausea (Gastrointestinal disorders) | 13 | 19
Vomiting (Gastrointestinal disorders) | 6 | 7
Chills (General disorders) | 3 | 4
Fatigue (General disorders) | 20 | 30
Fever (General disorders) | 5 | 6
Flu like symptoms (General disorders) | 2 | 0
Non-cardiac chest pain (General disorders) | 3 | 3
Pain (General disorders) | 8 | 11
Infections and infestations - Other (Infections and infestations) | 2 | 0
Lung infection (Infections and infestations) | 4 | 4
Urinary tract infection (Infections and infestations) | 3 | 2
Dermatitis radiation (Injury, poisoning and procedural complications) | 6 | 3
Alkaline phosphatase increased (Investigations) | 4 | 4
Creatinine increased (Investigations) | 2 | 2
Lymphocyte count decreased (Investigations) | 9 | 10
Lymphocyte count increased (Investigations) | 2 | 0
Neutrophil count decreased (Investigations) | 7 | 9
Platelet count decreased (Investigations) | 10 | 8
Weight loss (Investigations) | 6 | 11
White blood cell decreased (Investigations) | 12 | 12
Anorexia (Metabolism and nutrition disorders) | 13 | 11
Glucose intolerance (Metabolism and nutrition disorders) | 2 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 8 | 12
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 | 7
Hypocalcemia (Metabolism and nutrition disorders) | 4 | 8
Hypomagnesemia (Metabolism and nutrition disorders) | 4 | 9
Hyponatremia (Metabolism and nutrition disorders) | 4 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 3
Chest wall pain (Musculoskeletal and connective tissue disorders) | 6 | 2
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3 | 2
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 2 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 3
Dizziness (Nervous system disorders) | 6 | 5
Dysgeusia (Nervous system disorders) | 4 | 6
Headache (Nervous system disorders) | 4 | 5
Paresthesia (Nervous system disorders) | 4 | 3
Peripheral sensory neuropathy (Nervous system disorders) | 6 | 11
Anxiety (Psychiatric disorders) | 3 | 5
Depression (Psychiatric disorders) | 4 | 3
Insomnia (Psychiatric disorders) | 5 | 6
Urinary retention (Renal and urinary disorders) | 2 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 9 | 3
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 14
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 16 | 17
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 10 | 5
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 7 | 3
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Sore throat (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 6 | 12
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 | 13
Hypertension (Vascular disorders) | 2 | 1
Hypotension (Vascular disorders) | 4 | 3
Thromboembolic event (Vascular disorders) | 2 | 0

LIMITATIONS AND CAVEATS:
Following a recommendation on July 13, 2015 by the NRG Data Monitoring Committee accrual was halted early after accruing only 71 of 97 patients due to unexpectedly high rates of grade 5 toxicity on the panitumumab arm.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI's are required to abide by the sponsor's publication guidelines which require review by coauthors and subsequent review and approval by the sponsor.